CLINICAL TRIAL: NCT04185103
Title: Changes in the T-wave Alternans in Patients With Heart Failure Treated Wih Sacubitril-Valsartan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Agencia Sanitaria Bajo Guadalquivir (Unknown)
Responsible Party: Sponsor
Other Study IDs: FIS-SAC-2018-02
Record Dates: First submitted 2019-11-12; First posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Heart Failure
Keywords: Heart Failure; Sacubitril-Valsartan; T-wave changes alternans
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sacubitril-Valsartan cohort: Patients with left systolic disfunction (left ventricle ejection fraction<40%) heart failure and diagnosed with grade II heart failure that have been treated with an ACE or ARA II+betablocker at stable doses during the last 4 weeks and after being evaluated by the cardiologist start Sacubitril-Valsartan treatment.
  Interventions: Drug: Sacubitril-Valsartan

INTERVENTIONS:
Drug: Sacubitril-Valsartan — After signing the Informed Consent, in the shortest possible time, the study investigator will carry out an ergometric test for the T-wave alternans (TWA) while still taking the basal medication. The patient will also sign the prototype Informed Consent for carrying out a stress test on a treadmill. It will also be carried out a basal life quality questionnaire, an analytical determination and a colour doppler echocardiography.

SUMMARY:
The aim of this study is to know if the Sacubitril-Valsartan treatment improves the T-wave alternans in those patients that begin its treatment, which would indirectly show a lower risk of malignant ventricular arrythmias.

DETAILED DESCRIPTION:
Sacubitril-Valsartan has shown to reduce sudden death in its principal clinical trial, PARADIGM-HF.

A T wave alternans (TWA) is an electrophysiological phenomenon that acts as an independent predictor of sudden death and ventricular arrhythmias in postinfarct myocardial.

TWA is measured by using a special software and electrodes during a treadmill test, that analyse small changes in the microvolt of the T wave consecutive with a complex algorithm in three dimensions. The TWA could be negative (normal), positive (pathological) or indeterminate. If a TWA is pathological it reflects an electric instability in depolarization.

Our hypothesis is that the treatment with Sacubitril-Valsartan in heart failure patients with reduced ejection fraction, could improved the TWA.

ELIGIBILITY:
Inclusion Criteria:

* Adults from 18 to 80 years old.
* Patients with grade II heart failure according to the New York Heart Association (NYHA).
* Left systolic disfunction: left ventricle ejection fraction<40%
* NT-proBNP > 600 pg/ml (or > 100 pg/ml in the case the patients has been hospitalised during the last year.
* Treated with ACE or ARA II+betablocker at stable doses during the prior 4 weeks to the beginning of the study.

Exclusion Criteria:

* Previously treated with Sacubitril-Valsartan.
* Allergy or intolerance to ARA II.
* Systolic blood pressure < 100 mmHG at inclusion.
* Glomerular Filtration <35 ml / min / 1.73 m2 of body surface.
* Level of potassium > 5,4 mEq/l.
* Impossibility to walk on a treadmill.
* Record of recovered sudden death or documented ventricular tachycardia.
* Carrier of an automatic implantable defibrillator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with heart failure that meet all of the following criteria and none of the exclusion criteria.
  The selection of patients to be included in the study will be made in accordance to the Sacubitril-Valsartan data sheet.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-11-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Analyze the changes in the T-wave alternans | Up to 6 months after the beginning of the Sacubitril-Valsartan treatment
  Comparison of the results in the same patient just before the beginning of the Sacubitril-Valsartan pharmacological treatment versus 6 months after its beginning, in patients with grade II heart failure and left systolic disfunction (left ventricle ejection fraction<40%).

SECONDARY OUTCOMES:
Evaluate the results in the life quality questionnaire. | Up to 6 months after the beginning of the Sacubitril-Valsartan treatment
  Comparison of the life quality questionnaires results before and after the Sacubitril-Valsartan treatment.
Study the levels of the n-terminal type B natriuretic propeptide | Up to 6 months after the beginning of the Sacubitril-Valsartan treatment
  Comparison of the n-terminal type B natriuretic propeptide levels before and after the Sacubitril-Valsartan treatment.
Evaluate the echocardiographic results | Up to 6 months after the beginning of the Sacubitril-Valsartan treatment
  The echocardiographic results will be assessed by a combination of the measurement of the parameters: left ventricular ejection fraction (LVEF), left ventricular end-diastolic volume (LVEDV), left ventricular end systolic volume (LVESV) and left ventricle diastolic function, that will be compared before and after the Sacubitril-Valsartan treatment to evaluate its effect in patients with heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio José Fernández Romero, Dr, Principal Investigator — Hospital de Alta Resolución de Utrera; Antonio José Fernández Romero, Dr, Study Chair — Hospital de Alta Resolución de Utrera
Locations (4):
- Spain (4):
  - Hospital de Alta Resolución de Utrera, Utrera, Sevilla
  - Hospital de Alta Resolución de Sierra Norte, Constantina, Seville
  - Hospital de Alta Resolución de Écija, Écija, Seville
  - Hospital de Alta Resolución de Lebrija, Lebrija, Seville

IPD SHARING:
Plan to Share IPD: No